CLINICAL TRIAL: NCT02733783
Title: Design of a Model to Study Functionality of the Trigeminal Nerve in Relation to Controlled Nasal Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Garyafalia Lekakis, Research Associate, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S59058
Record Dates: First submitted 2016-03-17; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Fracture of Nasal Bones, Sequela

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- septorhinoplasty patients (Experimental): Elective septorhinoplasty patients that will undergo bilateral osteotomies. All the patients will undergo cold dry air provocation and 3 hours later capsaicin provocation, during a preoperative visit, one week before the intervention and during three post-operative visits two weeks, three months and six months.
  Interventions: Device: Cold dry air machine

INTERVENTIONS:
Device: Cold dry air machine — Cold Dry Air (CDA)- nasal provocation: Compressed dry air is delivered through a transparent anaesthesia mask placed over the nose and mouth of the patients. Subjects are instructed to breath through the nose only. Exposure to CDA lasts for 15 minutes. The flow, measured by a gas flow analyzer of Dräger was set at 12,5 l/min. The temperature of the air reaching the nose is at -10° C with a relative humidity of 10%-15%.

SUMMARY:
The primary aim of the study is to create a model; in order to examine the effects of neural trauma in patients that are healthy individuals, induced by controlled nasal fractures during rhinoplasty, and the regeneration process in the weeks/months that follow. This study includes monitoring of subjective nasal symptoms with a visual analogue scale (VAS) score, peak nasal inspiratory flow (PNIF) measurements, collection of nasal secretions and nasal provocation (response to capsaicin and cold dry air (CDA) exposure).

DETAILED DESCRIPTION:
The investigators will set up a prospective mono-center study. The investigators will utilize objective and subjective parameters in order to assess trigeminal nerve function at the level of the nasal mucosa before and after septorhinoplasty (as a model of controlled nasal fractures). The subjective parameters involve a visual analogue scale (VAS) score for each individual nasal symptom (nasal obstruction, facial pain/pressure, headache, rhinorrhea, sneezing, pruritus, post nasal drip, and loss of smell). An objective assessment includes measurement of PNIF (Peak Nasal Inspiratory Flow), the presence of neuropeptides in nasal secretions, (by introducing merocels and removing them 5 minutes later), short cold dry air (CDA) provocation and capsaicin provocation with subsequent measurements of PNIF and VAS scores and neuropeptides.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing septorhinoplasty, with planned bilateral osteotomies
2. No rhinological symptoms/complaints (rhinorrhea, sneezing, itchiness, nasal obstruction)
3. Age > 18 and < 65 years
4. Written informed consent
5. Willingness to adhere to visit schedules
6. Adequate contraceptive precautions in female patients with childbearing potential

Exclusion Criteria:

1. Age < 18 and > 65 years
2. Patients with nasal symptoms at baseline, defined as having more than 2,5 on VAS score

   for individual nasal symptoms related to mucosal pathology
3. Nasal endoscopic signs of inflammatory pathology (rhinitis, rhinosinusitis with/without

   nasal polyps)
4. Use of systemic steroid treatment, intranasal steroid treatment, oral leukotriene antagonists

   or long acting antihistamines?
5. Asthma
6. Pregnancy or breastfeeding
7. Any disorder of which might compromise the ability of a patient to give truly informed

   consent for participation in this study.
8. Enrollment in other investigational drug trial(s) or is receiving other investigational

   agent(s) for any other medical condition.
9. Contra-indications for local anaesthesia (Cocaine 5%)
10. Smoking
11. Systemic disease with lesions in ENT domain
12. Malignancies or severe comorbidity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
changes from baseline PNIF (peak nasal inspiratory flow) at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  Short Cold Dry Air (CDA) provocation with symptom evaluation using VAS and PNIF post-provocation and collection of nasal fluid by Merocel after provocation.
changes from baseline VAS (visual analogue score) for nasal obstruction at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of nasal obstruction will be evaluated on a VAS scoring system (0-10 cm) on the baseline visit and on follow-up visits. All patients will be asked to mark their nasal obstruction on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline level of neuro mediators in nasal secretions, at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  Collection of nasal fluid: nasal fluid will be collected, by placing a small Merocel (4 cm) between the middle and inferior turbinate, for 5 minutes. This technique is a traumatic and painless for the patient, and allows a rapid collection of nasal fluid without the need for local anesthesia. The fluid will be stored at -20°C until analysis, i.e. measurement of mediators such as histamine, Substance P (SP), Neurokinin A and B (NKA, NKB), Nerve Growth Factor (NGF), eotaxin, NPY, CGRP by ELISA. All these measurements will be aggregated to arrive at one reported value an increase of neuro mediators in the immediate postoperative period and gradual decrease to the baseline levels over a period of time.
changes from baseline VAS (visual analogue score) for rhinorrhea at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of rhinorrhea will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their nasal rhinorrhea on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline VAS (visual analogue score) for facial pain at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of facial pain will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their facial pain on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline VAS (visual analogue score) for sneezing at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of sneezing will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their sneezing on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of facial pain will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their facial pain on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of sneezing will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their sneezing on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline VAS (visual analogue score) for pruritus at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of pruritus will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their pruritus on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of pruritus will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their pruritus on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of sneezing will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their sneezing on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline VAS (visual analogue score) for catarrh at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of catarrh will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their catarrh on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of pruritus will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their pruritus on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of catarrh will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their catarrh on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline VAS (visual analogue score) for sense of smell at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of facial pain will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their facial pain on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of pruritus will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their pruritus on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of hyposmia will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their sense of smell on this VAS score on all visits before and after CDA and capsaicin provocation.
changes from baseline VAS (visual analogue score) for headache at 2 weeks, 3 and 6 months after rhinoplasty | Before and after each test (cold dry air provocation) during the pre-operative visit (one week before the intervention) and the three postoperative visits (two weeks, three months and six months after the intervention)
  The presence of facial pain will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their facial pain on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of pruritus will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their pruritus on this VAS score on all visits before and after CDA and capsaicin provocation.
  The presence of headache will be evaluated on a VAS scoring system (0-10 cm) on the baseline and follow-up visits. All patients will be asked to mark their headache on this VAS score on all visits before and after CDA and capsaicin provocation.